CLINICAL TRIAL: NCT00219934
Title: Observational Study of Treated and Untreated Acute and Early HIV-1 Infection
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: Aaron Diamond AIDS Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMA 0465
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infections
Keywords: New HIV Infection; Acute HIV Infection; Primary HIV Infection; Acute Seroconversion Syndrome
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PLASMA AND PERIPHERAL BLOOD MONONUCLEAR CELLS
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: acute or early in the course of HIV-1 infection, independent of decisions regarding therapy with HAART.
  Interventions: Drug: Antiretroviral therapy
- Group B: subjects who were diagnosed with acute HIV-1 infection in the past and have been participating in an ADARC/Rockefeller University Hospital treatment protocol for acute HIV-1 infection, and currently have a viral load consistently less than 50 copies/ml on current treatment
  Interventions: Drug: Antiretroviral therapy

INTERVENTIONS:
Drug: Antiretroviral therapy — HAART therapy

SUMMARY:
Group A: Long-term follow-up is needed for subjects identified as acute or early in the course of HIV-1 infection, independent of decisions regarding therapy with highly active anti-retroviral therapy (HAART).

Group B: This protocol will also be offered to subjects who were diagnosed with acute HIV-1 infection in the past and have been participating in an ADARC/Rockefeller University Hospital treatment protocol for acute HIV-1 infection, and currently have a viral load consistently less than 50 copies/ml on current treatment (Group B)

DETAILED DESCRIPTION:
At the initial visit: subjects will undergo a complete history and physical examination. They will have blood drawn for HIV-1 antibody testing, resistance testing, and lymphocyte subsets. In addition, blood will be drawn for hematology, chemistries, and syphilis, and Hepatitis B and C serologies.

Individuals in Group B will not have HIV-1 antibody testing, resistance testing, or Hepatitis B and C serologies performed, as these would have been performed as part of their current protocol. Individuals electing to initiate antiretroviral therapy will obtain standard HAART as prescribed by their physicians.

Group A subjects will be seen at Weeks 4, and 12 ,then every 12 weeks until week 48, then every 24 weeks until week 96. If treated during acute and early infection, then they will be seen every 48 weeks thereafter for 5 years. If untreated during acute and early infection, then they will be discontinued from the study.

Group B participants who have been followed for less than 96 weeks will be seen every 12 weeks until week 48, then every 24 weeks until week 96.

Participants currently enrolled beyond week 96 who were treated during acute and early infection, and whose treatment was uninterrupted, will be seen every 48 weeks. If participants were not treated during acute and early infection, or treatment was interrupted, then they will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Group A: HIV-1 infected individuals at least 16 years of age with HIV-1 RNA detectable in the blood (>2000 copies/ml) and one of the following:

  1. a negative test for HIV-1 antibodies
  2. an indeterminate test for HIV-1 antibodies
  3. a positive test for HIV-1 antibodies with an immature Western Blot (less than 5 bands) which subsequently matures (addition of 2 or more bands)
  4. a positive test for HIV-1 antibodies and a documented negative test within 6 months of presentation
  5. a positive test for HIV-1 antibodies with a simultaneous negative low sensitivity ("detuned") assay (S/C <15)
  6. Individuals must be able and willing to provide written informed consent

Group B: Approximately 90 individuals diagnosed with acute HIV-1 infection in the past who have been participating in an ADARC/Rockefeller University Hospital protocol involving treatment of acute HIV-1 infection and are currently on that regimen with HIV-1 RNA consistently less than 50 copies/ml and are interested in changing to a protease inhibitor-sparing regimen or may continue to be treated with medications provided or taken as part of a completed ADARC/RUH study of the treatment of acute and early HIV infection

Exclusion Criteria:

* Individuals less than 16 years of age
* Individuals who are unable or unwilling to provide written informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the community or from existing ADARC clinical trials. Participants will give written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2002-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Development of AIDS or AIDS-defining conditions as per the CDC | end of study
Death due to AIDS or AIDS-defining conditions | end of study
Morbidity due to therapy | end of study
Death due to therapy | end of study

SECONDARY OUTCOMES:
HIV-1 RNA levels | duration of the study
T-cell subsets | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- See also: The Aaron Diamond AIDS Research Center — http://www.adarc.org